CLINICAL TRIAL: NCT02374398
Title: A Randomized, Controlled Clinical Trial Comparing the Use of Intravenous Tranexamic Acid With Aquamantys Bipolar Sealer for Blood Loss Reduction in Primary Total Knee Arthroplasty
Brief Title: Clinical Trial Comparing Tranexamic Acid (TXA) With Aquamantys Sealer in Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eastern Maine Medical Center (Other)
Responsible Party: Principal Investigator, Alexandru Seviciu, MD, Anesthesiologist, Eastern Maine Medical Center
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 10-1-M-194
Record Dates: First submitted 2015-01-30; First posted 2015-02-27 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Blood Loss
Keywords: Tranexamic Acid; Blood Loss; Aquamantys System; TKA
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Tranexamic Acid (Active Comparator): TXA will be provided ready-to-use as IV infusion with instructions written by the pharmacy department. The TXA dose will be 20mg/kg to be administered as a bolus over 20 minutes
  Interventions: Drug: Tranexamic Acid
- Aquamantys System (Active Comparator): The Aquamantys system will be used as indicated by orthopedic surgeon intraoperative. Local temperatures under 100°C are sufficient to shrink collagen fibers in the walls of blood vessels, effectively sealing the blood vessels. Simultaneous RF power and saline delivery. Power settings from 20-200 watts
  Interventions: Device: Aquamantys System
- TXA plus Aquamantys (Active Comparator): TXA will be provided ready-to-use as IV infusion with instructions written by the pharmacy department. The TXA dose will be 20mg/kg to be administered as a bolus over 20 minutes.
  The Aquamantys system will be used as indicated by orthopedic surgeon intraoperative. Local temperatures under 100°C are sufficient to shrink collagen fibers in the walls of blood vessels, effectively sealing the blood vessels. Simultaneous RF power and saline delivery. Power settings from 20-200 watts.
  Interventions: Drug: Tranexamic Acid; Device: Aquamantys System
- Control (Placebo Comparator): Saline will be provided ready-to-use as IV infusion with instructions written by the pharmacy department. The saline dose will be administered as a bolus over 20 minutes
  Interventions: Other: Control

INTERVENTIONS:
Drug: Tranexamic Acid — see arm/group descriptions
  Other Names: Cyklokapron
  Arms: TXA plus Aquamantys; Tranexamic Acid
Device: Aquamantys System — see arm/group descriptions
  Arms: Aquamantys System; TXA plus Aquamantys
Other: Control — Standard Electro-cautery and Saline
  Other Names: Placebo
  Arms: Control

SUMMARY:
The aim of the study is to determine if the use of iv TXA or Aquamantys system improve the postoperative hemoglobin and hematocrit after primary TKA and what is the effect of the simultaneous use of iv TXA and Aquamantys on the postoperative hemoglobin and hematocrit. The assumption is that the combination of iv TXA and Aquamantys system will enable an improvement in the postoperative hemoglobin and hematocrit equal or larger than the improvement generated by the use of Aquamantys system alone.

DETAILED DESCRIPTION:
The study is randomized, placebo controlled. The study population includes patients older than 18 years of age undergoing elective total primary knee replacement under spinal anesthesia. All patients enrolled in the study will undergo TKA performed by the same orthopedic surgeon. Since controversies exist regarding the effect of different types of anesthesia (general anesthesia versus spinal or epidural anesthesia) on intraoperative blood loss, in order to eliminate an important confounding variable we decided to exclusively enroll for our study patients that qualify for and agree with spinal anesthesia to be used as the main anesthetic technique for their TKA.

All clinical trial procedures will be performed by personnel blinded to study treatment assignment. Unblinding is only allowed for safety concerns in an emergency situation.The only other exception is represented by the surgeon, who can't be blinded in regards to using Aquamantys system and the bipolar sealer. Once a subject becomes eligible for the trial, the investigator or the designee will access the randomization system.

Enrolled subjects will be assigned to one of the 4 groups by block randomization of alternating 4 and 8 and 12 patients per block. The Pharmacy Department will provide the iv placebo or the iv TXA according to the randomization process.

This clinical trial will be conducted in accordance to this protocol, Good Clinical Practice and applicable regulatory requirements

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over age of 18 undergoing elective total primary knee arthroplasty under spinal anesthesia.

Exclusion Criteria:

* Previous adverse reaction to tranexamic acid
* Congenital or acquired coagulation disorders
* Preoperative platelet count of less than 100,000/microliter or INR> 1.4
* History of deep venous thrombosis, pulmonary embolism or cerebrovascular accident
* Patients with acquired defective color vision
* Renal insufficiency (Glomerular filtration rate <20 ml/min)
* Severe liver disease
* Coronary stents
* Pregnant patients
* Main anesthetic other than spinal anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2011-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Sorondo, MD, Study Director — Eastern Maine Medical Center
Locations (1):
- Eastern Maine Medical Center, Bangor, Maine, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- TXA Plus Aquamantys: TXA will be provided ready-to-use as IV infusion with instructions written by the pharmacy department. The TXA dose will be 20mg/kg to be administered as a bolus over 20 minutes.
  The Aquamantys system will be used as indicated by orthopedic surgeon intraoperative. Local temperatures under 100°C are sufficient to shrink collagen fibers in the walls of blood vessels, effectively sealing the blood vessels. Simultaneous RF power and saline delivery. Power settings from 20-200 watts.
  Tranexamic Acid: see arm/group descriptions
  Aquamantys System: see arm/group descriptions
- Control: Saline will be provided ready-to-use as IV infusion with instructions written by the pharmacy department. The saline dose will be administered as a bolus over 20 minutes
  Control Group: Saline and Standard Elecdrocautery
Period: Overall Study
Arm/Group | Tranexamic Acid | Aquamantys System | TXA Plus Aquamantys | Control
Started | 31 | 32 | 32 | 32
Completed | 29 | 31 | 29 | 32
Not Completed | 2 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Aquamantys System | TXA Plus Aquamantys | Control | Total
Number analyzed (Participants) | 29 | 31 | 29 | 32 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (8.6) | 64.8 (8.0) | 61.1 (10.5) | 62.9 (8.4) | 63.6 (8.9)
Gender [Count of Participants; unit: Participants]
  Female | 15 | 17 | 16 | 18 | 66
  Male | 14 | 14 | 13 | 14 | 55
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 29 | 32 | 121

OUTCOME MEASURES:

1. Primary Outcome: The Change in Hemoglobin (Hb) From the Day of Surgery
Description: 1. Control group- iv placebo normal saline plus regular electrocautery.
  2. iv TXA plus regular electrocautery.
  3. iv placebo plus Aquamantys system and regular electrocautery.
  4. iv TXA and Aquamantys system and regular electrocautery
Time Frame: day of surgery preoperative time to postoperative day 3 or postoperative day 2 if day 3 data are not recorded for the 4 groups
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Tranexamic Acid | Aquamantys System | TXA Plus Aquamantys | Control
Number analyzed (Participants) | 29 | 31 | 29 | 32
g/dl | 2.6 (0.9) | 3.2 (1.1) | 2.6 (1.0) | 3.7 (1.1)

2. Primary Outcome: The Change in Hematocrit (Ht) From the Day of Surgery
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Volume % of RBC in blood
Arm/Group | Tranexamic Acid | Aquamantys System | TXA Plus Aquamantys | Control
Number analyzed (Participants) | 29 | 31 | 29 | 32
Volume % of RBC in blood | 7.1 (2.51) | 8.6 (3.22) | 6.8 (2.58) | 10.0 (3.38)

3. Secondary Outcome: Post Operative Blood Loss
Description: The estimated blood loss was determined with the Gross formula [23]. According to a review article published in 2013, Gross's formula though developed in 1983 is still widely used as reported. The formula which is relatively easy to use is described below:
  Patient blood volume (PBV) = K (1) x height (m) 3 + K (2) x weight (kg) + K (3) Where K (1) = 0.3669 (male), 0.3561(female); K (2) = 0.03219 (male), 0.03308 (female); And K (3) = 0.6041(male), 0.1833 (female) Estimated blood loss = PBV [Hematocritinitial - Hematocritfinal ] / Hematocritmean Where mean hematocrit is the sum of initial and final hematocrit divided by two.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Tranexamic Acid | Aquamantys System | TXA Plus Aquamantys | Control
Number analyzed (Participants) | 29 | 31 | 29 | 32
ml | 747.9 (298) | 938.9 (376) | 746.6 (270) | 1077.6 (371)

4. Secondary Outcome: Cost Analysis
Description: Charges per case.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Tranexamic Acid | Aquamantys System | TXA Plus Aquamantys | Control
Number analyzed (Participants) | 29 | 31 | 29 | 32
Dollars | NA (NA) — IRB censored | NA (NA) — IRB censored | NA (NA) — IRB censored | NA (NA) — IRB censored

5. Secondary Outcome: Adverse Events
Description: Complications: deep venous thrombosis(DVT) or arterial thrombosis, pulmonary embolism(PE), myocardial infarction (MI), cerebrovascular accident (CVA)
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid | Aquamantys System | TXA Plus Aquamantys | Control
Number analyzed (Participants) | 29 | 31 | 29 | 32
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Tranexamic Acid | Aquamantys System | TXA Plus Aquamantys | Control
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/31 | 0/32 | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes